CLINICAL TRIAL: NCT03304626
Title: A Pilot Study to Evaluate the Efficacy and Safety of Budesonide as an Alternative to Prednisone for Liver Transplant Immune Suppression
Brief Title: Budesonide for Liver Transplant Immune Suppression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: American College of Gastroenterology (Other)
Responsible Party: Principal Investigator, Khurram Bari, Assistant Professor, University of Cincinnati
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-1488
Record Dates: First submitted 2017-10-03; First posted 2017-10-09 (Actual); Results first posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-06

CONDITIONS: Acute Cellular Graft Rejection; New Onset Diabetes After Transplant
MeSH Terms: interventions — Budesonide; Prednisone

STUDY DESIGN:
Intervention Model Description: 20 subjects will receive open label Budesonide along with standard immune suppression and their outcomes will be compared to 20 matched controls receiving standard of care treatment including prednisone plus standard immune suppression
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Budesonide EC 3 mg capsule. The dose will be as follows
  Time post Liver Transplantation Immunosuppressive therapy Days 0-3 Standard immune suppression (SIS) + Intravenous corticosteroids Days 4-30 SIS + Budesonide 9 mg Days 31-45 SIS + Budesonide 6 mg Days 46-90 SIS + Budesonide 3 mg Days 90 onwards SIS1
  Interventions: Drug: Budesonide 3Mg Capsule
- Control Group (Active Comparator): Standard of Care
  Time post Liver Transplantation Immunosuppressive therapy Days 0-3 Standard immune suppression (SIS) + Intravenous corticosteroids Days 4-30 SIS + Prednisone 15-60 mg Days 31-45 SIS + Prednisone 10 mg Days 46-90 SIS + Prednisone 2.5 to 7.5 mg Days 90 onwards SIS
  Interventions: Drug: Standard of Care Prednisone

INTERVENTIONS:
Drug: Budesonide 3Mg Capsule — Budesonide capsule in place of prednisone (standard of care)
  Other Names: Entocort EC
  Arms: Study Group
Drug: Standard of Care Prednisone — Prednisone taper (Standard of Care)
  Other Names: Prednisone
  Arms: Control Group

SUMMARY:
This is a pilot study that investigates the efficacy and safety of budesonide as an immune suppressing agent for liver transplant recipients in the early post-transplant period.

The primary end-point is rates of acute cellular rejection within first 24 weeks post-liver transplant. Secondary end points include rates of new onset diabetes after transplant and safety of budesonide.

The study is structured as a prospective clinical trial. After receiving 4 days of intravenous corticosteroids on liver transplant post-operative days 0 through 3, subjects will be started on standard immunosuppression plus enteric coated budesonide (study drug) in place of standard immune suppression plus prednisone (standard of care). Study drug will be tapered over 12 weeks in accordance with the existing standard of care immune suppression protocol. Subjects will be followed in outpatient transplant clinic for 24 weeks. The purpose of the study is to conduct a pilot study to generate rates and effect size that can be used in a subsequent equivalent trial. A total of 20 subjects will be enrolled to receive the standard immunosuppression plus budesonide and their outcomes will be compared to 20 controls receiving standard immunosuppression plus prednisone (standard of care). The use of controls is to generate rate and variability that can be compared with the rate obtained from patients that receive study drug by examining the 95% confidence band.

DETAILED DESCRIPTION:
Enrollment of Subjects: All consecutive patients undergoing liver transplant (LT) at the University Of Cincinnati Transplant Center will be screened for enrollment upon admission for transplant surgery. Subjects will be approached after permission from attending on record by one of the members of research team. Study rationale, procedures, different interventions, potential benefits and risks as well as alternatives to study participation will be explained to the subjects in their native language in non-medical terms, as much possible. For non-English speakers, certified interpreter services will be used. Subjects meeting all of the inclusion and none of the exclusion criteria will be educated about the study and written informed consent will be obtained either 12 hours prior to undergoing LT or within 72 hours of completion of a successful transplant surgery. This time frame is proposed so that subjects have sufficient time to go over the study and are not pressured to sign the consent within a short time frame prior to LT surgery. In addition, all patients being placed on liver transplant list at our center will be provided with a copy of the consent form in the LT clinic at the time of listing for review only so that this study proposal is not completely novel to them at the time of LT surgery. A pregnancy test will be performed on all the females of childbearing potential.

Enrollment of Controls:

Each study subject will be matched with a control subject. Patients undergoing LT at University of Cincinnati that are not part of the study will serve as controls. Confounding and effect modifiers will be accounted for by matching the controls on multiple variables which may affect the primary outcome of ACR. These variables include: age less than 55 years, serum creatinine greater than 1.5 ng/mL, the use of antibody therapy at the time of transplant and a history of autoimmune hepatitis. To minimize the selection bias, the matched control will be selected in a manner that he/she would have undergone liver transplantation within a 24 week period (8 weeks prior or 16 weeks after) of the liver transplantation of the matched study subject. This means that data from controls will also be collected prospectively. Since outcomes are being measured at week 24 of liver transplantation, this will ensure that the investigators have no influence on selecting the controls with a known outcome. Controls will be identified through LT clinic. They will not undergo any study specific procedures, interventions, testing or evaluations. A written and informed consent will be obtained from all controls prior to their enrollment in the study. University of Cincinnati transplant program has performed 90-100 LTs each year over last 2 calendar years. Application of inclusion and exclusion criteria of our study to this database estimates that 65% of all LTs will be potential candidates for participation either as study subject or control. Based on this estimate the investigators are confident that this enrollment goal of 20 subjects and 20 controls can be achieved in 9-12 month period.

Study Drug:

After LT surgery, subjects will be started on SIS including intravenous corticosteroids, calcineurin inhibitor (CNI), mycophenolate mofetil (MMF) +/- thymoglobulin as per University of Cincinnati LT immune suppression protocol (UC-ISP).

On post-operative day 4, intravenous corticosteroids will be discontinued and replaced by the study drug; budesonide. Based on pharmacokinetic and bioavailability studies, 3 mg of budesonide is equivalent to 10 mg of prednisone. Starting dose of budesonide will be 9 mg by mouth daily which will be equivalent to 30-40 mg of prednisone used as standard of care. Study drug will be tapered over the next 3 months as detailed in Table 1 and in line with UC-ISP. At 3 months post LT, study drug will be discontinued. Subjects with autoimmune hepatitis as an etiology for LT will be initiated on prednisone 5 mg daily in addition to SIS as per UC-ISP.

Table 1: Study Drug Taper Time post Liver Transplantation Immunosuppressive therapy Days 0-3 Standard immune suppression (SIS) + Intravenous corticosteroids Days 4-30 SIS + Budesonide 9 mg Days 31-45 SIS + Budesonide 6 mg Days 46-90 SIS + Budesonide 3 mg Days 90 onwards SIS

Study Assessments (Visits 3-7):

Subjects will undergo study visits in the LT clinic or inpatient transplant unit at post-LT weeks 2,4,6,8 and 12 (Figure 1). At each visit, data regarding history and physical, vital signs, concomitant medications, use of hypoglycemic agents or insulin, adverse event assessment, laboratory blood work including blood counts, chemistries, blood glucose, liver function test, and tacrolimus trough level will be recorded. Blood samples for early morning cortisol level (between 6 AM and 9 AM) will be collected at week 4 and week 8 visits only. These samples will be centrifuged at 3600 rpm for 15 minutes, appropriately labelled and stored in - 80 C freezer at Schubert Research Clinic. All the samples from the study will be analyzed for serum cortisol in 1-2 batches to ensure uniform and standardized testing conditions and reagents. No other testing will be performed on these samples. Hemoglobin A1c will be checked at week 12 (visit 7). Additionally, at each visit, the study team will perform a pill count for the study drug. Study drugs will be dispensed every 4 weeks at study visits 2, 4 and 6. Decisions regarding obtaining a liver biopsy for evaluation of abnormal liver tests will be at the discretion of treating physician. Biopsy proven ACR will be treated according to UC-Rejection protocol.

Study drug will be discontinued at week 12 (visit 7) and subjects will continue routine post-LT follow up as per the current standard of care.

A low dose ACTH stimulation test will be performed at Schubert Research Clinic at week 12 visit. This test comprises of intravenous injection of cosyntropin at a dose of 1 micrograms per 1.73 m2 of body surface area and checking the serum cortisol levels at baseline and 30 minutes after cosyntropin injection. This test is used to assess adrenal insufficiency with a high sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subjects aged 21-75 years old
* Received a primary liver transplant within 4 days of enrollment

Exclusion Criteria:

* Received previous organ transplants
* Undergoing multiple organ transplants
* Recipients with advanced fibrosis in graft
* Treatment plan for subject includes receiving immunosuppressant therapy other than standard immune suppression (SIS) as per University of Cincinnati LT immune suppression protocol (UC-ISP).
* Inability to take enteral (orally or by tube feed) medications by day 4 post-transplant
* Subjects with diabetes mellitus prior to transplant (diabetes mellitus defined as use of hypoglycemic agents or HbA1c > 6.4 prior to transplant)
* Subjects who have any severe medical condition requiring acute or chronic treatment that in the investigator's opinion would interfere with study participation.
* Subjects who have been exposed to an investigational therapy within 30 days prior to enrollment or 5 half-lives on the investigational product, whichever is greater.
* Subjects in which concomitant use of medications which are inhibitors of CYP3A4 (such as ketoconazole, itraconazole, ritonavir, indinavir, saquinavir, erythromycin) cannot be avoided during the study period.
* Pregnant females
* Diminished mental capacity to consent for the study as determined by attending on the record.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Group: Budesonide EC 3 mg capsule. The dose will be as follows
  Time post Liver Transplantation Immunosuppressive therapy Days 0-3 Standard immune suppression (SIS) + Intravenous corticosteroids Days 4-30 SIS + Budesonide 9 mg Days 31-45 SIS + Budesonide 6 mg Days 46-90 SIS + Budesonide 3 mg Days 90 onwards SIS1
  Budesonide 3Mg Capsule: Budesonide capsule in place of prednisone (standard of care)
- Control Group: Standard of Care Controls that received
  Time post Liver Transplantation Immunosuppressive therapy Days 0-3 Standard immune suppression (SIS) + Intravenous corticosteroids Days 4-30 SIS + Prednisone 15-60 mg Days 31-45 SIS + Prednisone 10 mg Days 46-90 SIS + Prednisone 2.5 to 7.5 mg Days 90 onwards SIS
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control Group: Time post Liver Transplantation Immunosuppressive therapy Days 0-3 Standard immune suppression (SIS) + Intravenous corticosteroids Days 4-30 SIS + Prednisone 15-60 mg Days 31-45 SIS + Prednisone 10 mg Days 46-90 SIS + Prednisone 2.5 to 7.5 mg Days 90 onwards SIS
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [42 to 64] | 56 [44 to 63] | 56 [43 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 13 | 13 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 17 | 17 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Cellular Rejection Between Study and Control Groups
Description: Acute Cellular Rejection of liver graft was determined by liver biopsy using Banff criteria. The decision to perform liver biopsy was as per treating physician based on patient's clinical course and blood chemisteries. Protocol bioopsies were not performed.
Time Frame: Post-Transplant day 4 to week 24
Measure: Count of Participants; unit: Participants
Groups:
- Control Group: Standard of Care
  Time post Liver Transplantation Immunosuppressive therapy Days 0-3 Standard immune suppression (SIS) + Intravenous corticosteroids Days 4-30 SIS + Prednisone 15-60 mg Days 31-45 SIS + Prednisone 10 mg Days 46-90 SIS + Prednisone 2.5 to 7.5 mg Days 90 onwards SIS
  Standard of Care Prednisone: Prednisone taper (Standard of Care)
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 20 | 20
Participants | 1 | 1

2. Secondary Outcome: Rate of New Onset Diabetes After Transplant
Description: Rates of new onset diabetes in patients who did not have diabetes prior to liver transplant
Time Frame: Post-Transplant day 4 to week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 20 | 20
Participants | 0 | 3

3. Secondary Outcome: Number of Participants With Adrenal Suppression
Description: This outcomes was measured in Budesonide group only. Serum cortisol levels after 12 weeks of Budesonide use were checked to see if they fall below the adrenal suppression threshold of 3microgram/dl. If these were below 3 microgram/dl then patient is considered to have developed adrenal suppression.
  Second measure used to check for adrenal suppression was Cosyntorpin stimulation test. One-time, low-dose, cosyntropin stimulation test at week 12 was performed by administering cosyntropin at a dose of 0.5 µg/1.73 m2 of the body surface area and checking the serum cortisol levels at baseline and at 30 minutes after cosyntropin injection. A serum cortisol value of <11 µg/dL after cosyntropin stimulation was used to define adrenal suppression. Participant meeting any of these criteria was said to have developed adrenal suppression
Time Frame: Post-Transplant week 12
Population: This outcome was measured in study group only due to limited size and budget of the study
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 15 | 0
Participants | 2 |

4. Secondary Outcome: Number of Participants With Adverse Events
Description: Rates of adverse events
  1. All cause mortality
  2. Graft failure
  3. Acute cellular rejection
  4. New Onset Diabetes after Transplant
  5. Rates of bacterial, fungal or viral infections
  6. Other adverse events including ascites, pleural effusion, kidney injury, biliary stricture
Time Frame: Post-Transplant day 4 to week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 20 | 20
Participants | 10 | 6

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events recorded in Standard of Care Control Arm were limited to
  1. All cause mortality
  2. Graft failure
  3. Acute cellular rejection
  4. New Onset Diabetes after Transplant
  5. Rates of bacterial, fungal or viral infections
Arm/Group | Study Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 10/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=20) | Control Group (N=20)
Acute Kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0)
Ascites or Pleural effusion (Gastrointestinal disorders) | 3 (3) | 0 (0)
Bile leak (Gastrointestinal disorders) | 1 (1) | 0 (0)
Biliary stricture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=20) | Control Group (N=20)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-25): https://cdn.clinicaltrials.gov/large-docs/26/NCT03304626/Prot_SAP_001.pdf